CLINICAL TRIAL: NCT01136213
Title: Morphological and Functional Investigation of the Serotoninergic System in Multiple System Atrophy: a 18F-MPPF PET Study
Brief Title: Investigation of the Serotoninergic System in Multiple System Atrophy: a Positron Emission Tomography (PET) Study
Acronym: SEROTAMS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2008/01
Record Dates: First submitted 2010-05-26; First posted 2010-06-03 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Magnetic Resonance Spectroscopy; Fluoxetine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Multiple system atrophy
  Interventions: Radiation: PET (Positron Emission Tomography) Study; Other: Brain MRI (magnetic resonance imaging); Drug: Fluoxétine / Placebo
- Idiopathic Parkinson Disease
  Interventions: Radiation: PET (Positron Emission Tomography) Study; Other: Brain MRI (magnetic resonance imaging); Drug: Fluoxétine / Placebo
- Volunteers without neuropsychiatric disorder (Control)
  Interventions: Radiation: PET (Positron Emission Tomography) Study; Other: Brain MRI (magnetic resonance imaging); Drug: Fluoxétine / Placebo

INTERVENTIONS:
Radiation: PET (Positron Emission Tomography) Study — 5-HT1a auto-receptors will be visualized in vivo using 18F-MPPF PET study. Two PET studies will be performed, one after the intake of a single oral dose of fluoxetine and the other after placebo. The order of fluoxetine and placebo intake will be randomly assigned.
Other: Brain MRI (magnetic resonance imaging) — A brain MRI (magnetic resonance imaging)will be performed the day of the first PET study.
Drug: Fluoxétine / Placebo — The two PET studies will be performed, one after the intake of a single oral dose of fluoxetine and the other after placebo. The order of fluoxetine and placebo intake will be randomly assigned.

SUMMARY:
Multiple system atrophy (MSA) is a sporadic neurodegenerative disorder of the adult associated to a poor prognosis. MSA is clinically characterized by the association of extra-pyramidal, dysautonomic, cerebellar and pyramidal symptoms. Histological and biological studies have raised the hypothesis that, beside the well known dopamine deficiency, some of the symptoms could be related to a dysfunction in serotoninergic neurotransmission. Serotonin is involved in the modulation of several functions impaired in MSA, such as mood, motricity or sleep. The recent description of an association between loss of brainstem serotonin neurons and sudden death in patients with MSA reinforced the hypothesis of a critical role played by this neurotransmitter in the pathophysiology of this disease. Autoreceptors called 5-HT1a are strongly involved in the regulation of serotonin neurotransmission. During the last years several radio-ligands allowing in vivo PET quantification of 5-HT1a receptors, such as 18F-MPPF (4-(2'-methoxyphenyl)-1-[2'-(N-2''-piridinyl)-p-fluorobenzamide]methylpiperazine), were developed. Moreover, the investigators recently demonstrated the ability of this brain functional imaging method to investigate, in healthy volunteers, the functional properties of 5-HT1a autoreceptors through an evaluation of their desensitization after a single oral dose of fluoxetine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Multiple system atrophy (MSA)

  * MSA possible or probable
  * Male and female
  * Age : 30 to 80
  * No cognitive impairment
  * Unmodified treatment for 2 months
  * Able to give informed consent
  * Affiliated to social insurance
* Patients with idiopathic Parkinson's disease (IPD):

  * Positive clinical criteria for IPD
  * Male and female
  * Age : 30 to 80
  * No cognitive impairment
  * Unmodified treatment for 2 months
  * Able to give informed consent
  * Affiliated to social insurance
* Healthy controls:

  * Absence of neuropsychiatric disorder
  * Male and female
  * Age : 30 to 80
  * Able to give informed consent
  * Affiliated to social insurance

Exclusion Criteria:

* Patients with Multiple system atrophy (MSA)

  * Other Parkinsonian syndrome
  * Dementia
  * Recent intake (< 4 weeks or 8 weeks for fluoxetine) of medication acting on 5-HT1a receptors
  * History of major depression
  * Contraindication to brain MRI
  * Contraindication to PET
* Patients with idiopathic Parkinson's disease

  * Other Parkinsonian syndrome
  * Dementia
  * Recent intake (< 4 weeks or 8 weeks for fluoxetine) of medication acting on 5-HT1a receptors
  * History of major depression
  * Contraindication to brain MRI
  * Contraindication to PET
* Healthy controls:

  * Patient having a neuropsychiatric disease
  * Recent intake (< 4 weeks or 8 weeks for fluoxetine) of medication acting on 5-HT1a receptors
  * History of major depression
  * Contraindication to brain MRI
  * Contraindication to PET

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited by neurologists specialized in movement disorders
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
18F-MPPF binding potential - Biding potential (BP) under placebo in the raphe nucleus | Second visit (day 1)
  Amount of 5-HT1a autoreceptors (evaluated by measurement of 18F-MPPF binding potential) after intake of placebo in the raphe nucleus.

SECONDARY OUTCOMES:
18F-MPPF binding potential - Biding potential (BP) in other brain areas | Second visit (day 1)
  Amount of 5-HT1a autoreceptors (evaluated by measurement of 18F-MPPF binding potential) in other brain areas (brainstem, hippocampus, etc.)
Clinical parameters (motor handicap, orthostatic hypotension, quality of life, sleep, pain, tiredness) | Second visit (day 1)
18F-MPPF binding potential - Biding potential (BP) under placebo in other brain areas | Third visit (day 30)
  Amount of 5-HT1a autoreceptors (evaluated by measurement of 18F-MPPF binding potential) after intake of placebo in other brain areas (brainstem, hippocampus, etc.).
18F-MPPF binding potential - BP under fluoxetine in all brain areas | Third visit (day 30)
  Amount of 5-HT1a autoreceptors (evaluated by measurement of 18F-MPPF binding potential - BP) after intake of fluoxetine in all brain areas.
Clinical parameters (motor handicap, orthostatic hypotension, quality of life, sleep, pain, tiredness) | Third visit (day 30)

CONTACTS AND LOCATIONS:
Overall Officials: Igor SIBON, Pr, Principal Investigator — University Hospital Bordeaux (France); Geneviève CHENE, Pr, Study Chair — University Hospital Bordeaux (France)
Locations (3):
- France (3):
  - CHU de Bordeaux, Bordeaux
  - CHU Limoges, Limoges
  - CHU de Toulouse, Toulouse